CLINICAL TRIAL: NCT03796936
Title: Clinical Trial of 3MDR to Treat PTSD With mTBI, With and Without Eye Movement (3MDR)
Brief Title: 3MDR to Treat PTSD With mTBI (3MDR)
Acronym: 3MDR
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Walter Reed National Military Medical Center (U.S. Federal Agency)
Collaborators: Uniformed Services University of the Health Sciences (U.S. Federal Agency)
Responsible Party: Principal Investigator, Michael Roy, Professor of Medicine & Director, Division of Military Internal Medicine, Walter Reed National Military Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: WRNMMC-2018-0201
Record Dates: First submitted 2019-01-03; First posted 2019-01-08 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-07

CONDITIONS: Posttraumatic Stress Disorder; Traumatic Brain Injury
Keywords: posttraumatic stress disorder; traumatic brain injury; virtual reality; eye movement desensitization and reprocessing
MeSH Terms: conditions — Stress Disorders, Post-Traumatic; Brain Injuries, Traumatic | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This is a pilot, controlled clinical trial in which all 20 participants with comorbid PTSD and mTBI receive 10 sessions (3 preparatory, 6 3MDR treatment, and 1 conclusion), but will be randomized to either include eye movement, EM (EM+), or not (EM-).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- 3MDR With Eye Movement Component (EM+) (Experimental): All participants will complete 10 treatment sessions (3 preparatory, 6 3MDR and 1 concluding), led by a trained therapist, with the only difference between the intervention groups being the presence (EM+) or absence (EM-) of the eye movement component. For those in the EM+ intervention group, the EM component starts after the participant has thoroughly discussed a picture with the therapist; a red ball starts at one edge of the screen, moves rapidly back and forth across it, and upon reaching either edge, a 2-digit number appears superimposed in white on the ball. The number changes every time the ball meets either edge. The participant is asked to track the ball and call out the displayed numbers.
  Interventions: Behavioral: Motion-assisted, Multi-modular Memory Desensitization and Reconsolidation (3MDR) Therapy
- 3MDR Without Eye Movement Component (EM-) (Active Comparator): All participants will complete 10 treatment sessions (three preparatory sessions, six 3MDR sessions and one concluding session; see Table 1), led by a therapist who has been completed training in the conduct of this form of therapy, with the only difference between the intervention groups being the presence (EM+) or absence (EM-) of the eye movement component.There will be no exposure to the distractor stimulus (red ball) for those in the EM- intervention group.
  Interventions: Behavioral: Motion-assisted, Multi-modular Memory Desensitization and Reconsolidation (3MDR) Therapy

INTERVENTIONS:
Behavioral: Motion-assisted, Multi-modular Memory Desensitization and Reconsolidation (3MDR) Therapy — a novel treatment for PTSD combining aspects of virtual reality exposure therapy (VRET) and Eye Movement Desensitization and Reprocessing (EMDR), within the Computer Assisted Rehabilitation Environment (CAREN)

SUMMARY:
Background and Purpose: Posttraumatic stress disorder (PTSD) and mild traumatic brain injury (mTBI) are persistent and frequently comorbid complications of recent combat. There is no proven treatment for mTBI, and standard treatments for PTSD frequently achieve only transient, modest impact. Motion-assisted, Multi-modular Memory Desensitization and Reconsolidation (3MDR) is a novel treatment for PTSD combining aspects of virtual reality exposure therapy (VRET) and Eye Movement Desensitization and Reprocessing (EMDR), within the Computer Assisted Rehabilitation Environment (CAREN). The added benefit of the eye movement (EM) component of EMDR is controversial; the purpose of this pilot study is therefore to: 1) obtain an initial estimate of the efficacy of 3MDR in service members with comorbid PTSD and mTBI, and 2) determine the impact of EM on treatment response. The investigators hypothesize that 3MDR will significantly improve symptom severity, both with and without EM.

Population: Participants will be active or retired service members with a history of mTBI who meet criteria for probable PTSD on the PCL5. It is anticipated that participants will be recruited through the Center for Neuroscience and Regenerative Medicine (CNRM) Recruitment Core and the National Intrepid Center of Excellence (NICoE).

Design type and procedures: This is a pilot, controlled clinical trial in which all 20 participants with comorbid PTSD and mTBI receive 10 sessions (3 preparatory, 6 3MDR treatment, and 1 conclusion), but will be randomized to either include EM (EM+) or not (EM-). In the preparatory sessions, the therapist will help each participant select 2 songs and 14 pictures to be used in their treatment sessions. The therapist will help the participant rate the pictures from least to most impactful. Each 3MDR treatment session will start by playing the first song, to bring them back to the time of their trauma. This will be done while the participant walks on the CAREN's embedded treadmill through the 3MDR virtual environment (VE) projected onto the system's curved screen. This is followed by a display of one of their pictures, a manifestation of their trauma, which they directly face and walk down a hallway toward, until the picture looms before them. The therapist, standing next to the participant along the treadmill's edge, will query the participant about what the picture means to them, how it makes them feel, etc., while the CAREN operator superimposes key words (said by the participant) over the picture, which the therapist later asks the participant to read aloud. Then, for ~60 seconds, the EM+ group will see a red ball "bounce" across the screen in front of the picture, and a number appears on the ball as it touches the screen's edge. The participant will be asked to recite each number aloud. This element is absent for EM- participants. All participants repeats these procedures for 5-7 pictures in each 3MDR treatment session; the pictures used will be agreed upon by therapist and participant, targeting more impactful pictures, whether repeats or new, in later sessions. The pictures are followed by playing the second song, chosen to bring the participant back to present day. The participant will walk at a comfortable pace throughout the session, with each session lasting typically ~60 minutes. The primary outcome measure will be change in PCL-5 score from pre- to post-intervention, with additional measures at 3 and 6 months.

DETAILED DESCRIPTION:
This is a pilot prospective, randomized, interventional controlled clinical trial. Our study at the NICoE site will specifically target active or retired SMs who are OIF/OEF/OND veterans of any age and either gender who meet criteria for PTSD and have a lifetime history of mTBI. Comorbid PTSD and mTBI is highly prevalent in SMs and veterans of the recent wars in Afghanistan and Iraq, and having both diagnoses is associated with significantly greater symptom severity than either PTSD or mTBI alone (Brenner et al., 2010). TBI, the great majority of which is mTBI, is one of the most challenging, significant, and costly problems facing the DoD, and inhibiting readiness, whether in times of war or peace. Currently, no therapy has yet been proven efficacious in reducing persistent symptoms after TBI. Many patients with PTSD, particularly when it is combat-related, still suffer from substantial residual symptoms even after undergoing evidence-based psychotherapy (Watts et al., 2013; Bradley et al., 2001; Bison et al., 2007) and many even maintain their PTSD diagnosis (Steenkamp et al., 2015). The novel elements of 3MDR may prove to be particularly beneficial for those with both PTSD and a history of mTBI. If our approach is proven effective, there will be a sizeable population for whom this treatment could be provided, translating into both individual and DoD-wide benefit. Both TBI and PTSD have become signature wounds of the wars in Iraq and Afghanistan and pose significant health concerns for many military personnel. Currently, no intervention has yet been proven efficacious in reducing long-term symptoms of TBI. Furthermore, individuals with PTSD often have persistent symptoms even after completing validated treatments.

The proposed research has the potential to have a significant positive impact on the care of individuals with both PTSD and mTBI. As previously stated, 3MDR combines emotional exposure, dual-task processing, attenuation of working memory resources, and physical activity. Physical activity may be particularly beneficial in enhancing blood flow to the brain and facilitating production of beneficial factors such as brain-derived neurotrophic factor (BDNF). In addition, participants have the opportunity to demonstrate to themselves that they can actively overcome their avoidance by approaching and walking toward, or deliberately confronting, representations of their own traumatic memories. This approach may be particularly useful or of interest to veterans and SMs, who are accustomed to being physically active, may be less inclined to turn to pharmacotherapy than others with PTSD, and also have had high dropout rates and greater resistance to established, more traditional therapies. This relatively short treatment approach could have tremendous implications for improvement in symptoms as well as quality of life in individuals with PTSD and mTBI. Prior to any other study procedures, written informed consent will be obtained from each participant by the principal investigator (PI) or another study staff member trained by the PI to obtain informed consent. The PI will then complete a medical history and a series of questionnaires, to include a review of inclusion and exclusion criteria, to ensure that each participant is eligible to be enrolled in the study. A random number table will be used to randomly assign participants to either the eye movement (EM+) or no eye movement (EM-) group.

Table 1

Weeks Months 0

1 2 3 4 5 6 7 8 9 10 3 6 Consent X

3MDR Preparatory Sessions

X X X

3MDR CAREN Sessions

X X X X X X

Wrap-up Session

X

Post-Therapy Follow-Up

X X

Intervention All participants will complete 10 treatment sessions (three preparatory sessions, six 3MDR sessions and one concluding session; see Table 1), led by a therapist who has been completed training in the conduct of this form of therapy, with the only difference between the intervention groups being the presence (EM+) or absence (EM-) of the eye movement component. Dr. Eric Vermetten, head of research at the Military Mental Health unit of the Netherlands Ministry of Defense, and one of the developers of the 3MDR system, will conduct the training of all study therapists, will ensure that they are fully prepared to carry out the treatment protocol using the study manual he wrote, and he will provide regular supervision for the study therapists throughout the conduct of the study.

Preparatory Session 1: Research personnel will explain the upcoming 3MDR therapy sessions. Participants will be asked to identify 14 photographs, as well as two songs. The photographs may be digital, hard copy, or downloaded from the internet, and should be related to or reminiscent of the participant's traumatic experience. Each of the two songs are selected for specific purposes and will be played in their entirety during each of the 3MDR sessions. The first song is intended to bring them back to the time in which the trauma occurred; for example, for a service member with combat-related PTSD, this might be a song that they listened to a lot during their deployment. This will be played at the start of the 3MDR session while the participant walks at a comfortable pace through a virtual environment, before any of their pictures are displayed. The second song, on the other hand, is specifically chosen in order to bring them back to the present time, to remind them they are safe and are in the present moment.

Preparatory Session 2: The participant will share their photographs and music selections with the therapist. If the participant has difficulty identifying a sufficient number of appropriate photographs, the therapist will work with the participant during this session to identify why they may not have been able to come up with a sufficient number, and to help them find suitable options. This could include conducting online searches for publicly available pictures, including such options as Google Maps images of the area in which their trauma occurred. Sometimes, difficulty in the selection of pictures is a manifestation of the avoidance of any reminders of the traumatic, which is a cardinal feature of PTSD. The therapist may at this time explore the avoidance, if it is perceived to be a significant factor, and help the participant to work through and overcome it to a sufficient degree to identify suitable pictures to use in the treatment sessions. While the selection of songs does not usually pose as significant a challenge, the therapist will also review the participant's song selections, discuss why they were chosen, and try to ensure that the songs selected are suitable to take the participant back to the trauma, and then bring them back to the present and help them differentiate past from present, respectively. The therapist will then guide the participant to arrange their photographs according to their subjective units of distress (SUDS; Wolp,1969). The SUDS is a verbal self-report rating of subjective distress on a scale from 0-10, with 0 indicating no distress, and 10 representing maximum distress. The SUDS scale will be explained verbally to the participant and is not given via pencil and paper format. This will be used to rank the pictures for use during 3MDR treatment.

Preparatory Session 3: Participants will be introduced to, and familiarized with, the CAREN system (e.g., standing, shifting weight, and walking) located at the National Intrepid Center of Excellence (NICoE). Participants will be fitted by the engineer with a safety harness that will be worn for the entirety of each session that a participant is on the CAREN platform. In this session, a series of introductory applications will be used to familiarize the participant with the CAREN, which will take less than five minutes to perform. A short practice 3MDR session with a non-affecting photograph (e.g., a flower) will be conducted.

3MDR Sessions 1-6: A 3MDR trained therapist, as well as a CAREN engineer, will be present at every 3MDR therapy session.

Since sessions only include level treadmill walking, the platform will be disengaged with the bridge extended, as opposed to being separated from the main floor and set up to enable left-right and forward-backward shifts from the horizontal. This will minimize equipment noise and facilitate the communication between the therapist and participant. For participant monitoring and objective data collection, heart rate and kinematic data will be collected. A chest strap heart rate monitor will be worn by the participant throughout the session (Polar Electro Inc., Woodbury, NY; Zephyr Performance Systems, Annapolis, MD). Reflective motion capture markers will be placed on the participant's head, torso, and legs to measure biomechanics collected via motion capture cameras (Motion Analysis Inc., Santa Rosa, CA) that surround the CAREN.

Participants will then be fitted with an adjustable safety harness that fits comfortably over the shoulders. There is a risk of skin chafing if there is a lot of movement and the harness is not fitted properly. Each participant will be asked if they are comfortable throughout the study to mitigate this risk. The safety harness will be slipped into the safety support on the CAREN, which allows the participant to walk freely on the treadmill, but it does not allow them to walk off the platform. There is also a safety bar in front of the participant. The therapist will stand next to the participant during the session, on the edge of the platform but not on the treadmill. Up to seven pictures will be selected based on the participant's SUDS scores and/or themes agreed upon for each session. Pictures may be repeated during a session, reducing the number of pictures used for some sessions; this will be at the discretion of the treating therapist.

Each session has three phases: warm-up, intervention, and cool-down. The participant's preferred walking speed will be used to start the warm-up phase (2-5 min) and can be adjusted as needed. During this phase, the participant will virtually walk along an outdoor pathway toward a door while their chosen opening song plays to bring them back to a time of their trigger, as verbal guidance from their therapist prepares them for the intervention phase.

The CAREN system will be operated by a Biomedical Engineer, Sarah Kruger, who has been operating CAREN systems since 2007, and is certified by Motekforce Link. Motekforce Link is the manufacturer of the CAREN system. Motekforce Link provides CAREN operators with training and also verifies competencies required for system operation.

During utilization, the system is operated by a certified CAREN Operator and per protocol, at no time will the system be operated with less than two staff members in the room.

System checks are run daily by the CAREN Operator. All equipment is calibrated and maintained. Personnel from Motekforce Link visit annually to verify that everything is working properly and make any changes that are necessary.

In the intervention phase (50-55 min), the participant passes through an initial hallway leading to an open door that in turn leads them down a second hallway to approach their first picture, while being guided by the therapist with regard to what to do at each stage. The picture appears in the distance, but gradually becomes larger as they get closer to it, until it fills their field of vision. As soon as the participant is able to see the picture clearly, the therapist will request that they provide a detailed description of what the picture represents to them, and will then go on to ask the participant about their related memories and feelings. The therapist will verbally repeat key feelings and phrases that seem to carry particular meaning and resonance for the participant, so the CAREN engineer can type these words into the computer to have them appear superimposed over the picture (stage 1).

For those in the EM+ intervention group, the EM component will start after the participant has confirmed there are no more new feelings or words to be identified with the picture, and the therapist has asked the participant to read each of these words aloud, after which the engineer will remove the words from the screen but retain the picture. At this point a red ball will start at the left edge of the screen, and will move across the screen fairly rapidly from left to right, and upon reaching the right edge of the screen, a 2-digit number will appear superimposed on the red ball in white font (stage 2). The ball will then reverse course, passing from right to left, and the number will change as the ball meets the opposite edge of the screen. The ball will continue to move back and forth and the number will change every time the ball meets either edge of the screen. The participant will be asked to track the ball and call out the numbers displayed on the ball. After approximately 60 seconds, the distractor stimulus (ball image) is removed and a SUDS score is reported by the participant and recorded by the CAREN operator (stage 3). The participant will then walk out of the virtual hallway and onto an outdoor pathway that will lead them to another set of hallways, leading in turn to another picture, and the stages are repeated. There will be no exposure to the distractor stimulus (red ball) for those in the EM- intervention group.

After the last picture, the final phase of treatment (cool-down) begins (2-5 min). The session concludes with a piece of music, chosen by the participant to bring them back to the present time, typically a current favorite song of theirs. This music will be used to assist the participant in returning back to the present moment, while the therapist simultaneously provides them with positive feedback regarding their performance during the session, with a goal of achieving a significantly reduced SUDS score, which is reassessed at the end of the song.

Following the session, the CAREN operator will remove the safety harness from the participant. Participants will also be able to stop the session at any time if they feel ill or any motion sickness. A therapist-led discussion (approximately 15 minutes) with the participant will then occur in a private room; open questions will be used to elicit how the session was for the participant, and to discuss the purpose of re-experiencing to the participant in this setting. Notes made by the therapist will be stored, identified by study code and session number only, stored in password-protected files on a CAC-requiring computer. The study therapist will ensure the participant has completely returned to the present moment, has a reduced SUDS, and has ideally been able to attach a positive meaning to the 3MDR session. Participants will be asked to write their experiences and reflections down following each session in a diary format. All sessions will be recorded and a report summarizing the behavioral response to the intervention will be produced.

Concluding Session: Participants will provide their perception of how beneficial the treatment was, and if the current state of their symptoms will be discussed, with a focus on to what degree they have or have not improved compared to prior to their participation in the study.

Participants will return to the laboratory to complete follow-up assessments at 3 and 6 months. If participants are unable to return to the laboratory (i.e., no longer in the area), they will be contacted via phone, and the study questionnaires will be completed telephonically.

ELIGIBILITY:
Inclusion Criteria:

1. Military service member or veteran
2. Diagnosis of probable PTSD, as manifest by a PCL-5 score of 34 or greater
3. History of mild traumatic injury (mTBI) at least 3 months prior, documented by the OSU TBI-ID.

Exclusion Criteria:

1. History of moderate, severe, or penetrating TBI
2. History of a psychotic disorder, bipolar disorder, or active suicidal or homicidal ideation
3. Use of benzodiazepines on a regular basis within the past 30 days.
4. Inability to walk continuously, at a normal pace, for up to 60 minutes
5. Inability to follow verbal command and/or observe safety precautions
6. Women who are pregnant, based on self-reported date of last menses
7. Does not demonstrate capacity for informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — we seek to enroll 50% male, 50% female participants
Enrollment: 20 (Actual)
Dates: Start 2019-01-11 (Actual); Primary Completion 2022-01-22 (Actual); Study Completion 2022-06-22 (Actual)

PRIMARY OUTCOMES:
Change in PTSD Checklist for DSM5 (PCL-5) score | Post-intervention session 10, as well as 3 and 6 months later, compared to baseline
  The well-validated PCL-5 will assess self-reported PTSD symptom severity; range 0-84, higher score represents greater severity.

SECONDARY OUTCOMES:
Change in Neurobehavioral Symptom Inventory (NSI) score | Post-intervention session, and 3 and 6 months later, compared to baseline
  measure of postconcussive symptom severity; range 0-88, higher score represents greater severity
Change in Patient Health Questionnaire depression module (PHQ-9) score | Post-intervention session 10, as well as pre-intervention session 7, and 3 and 6 months later, compared to baseline
  measure of depression symptom severity; range 0-27, higher score represents greater severity
Change in Insomnia Severity Index (ISI) score | Post-intervention session 10, as well as pre-intervention session 7, 3 and 6 months later, compared to baseline
  measure of insomnia and sleep concerns; range 0-28, higher score represents greater severity

CONTACTS AND LOCATIONS:
Locations (1):
- Walter Reed National Military Medical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available via the Federal Interagency TBI Registry (FITBIR) after the study has been completed and all links to personal identifying information have been destroyed.
Supporting Information: CSR
Time Frame: Data will be made available after the completion of the study and destruction of links to personal identifying information, and then will be available indefinitely.
URL: https://fitbir.nih.gov/

REFERENCES:
- [Background] Roy MJ, Bellini P, Kruger S, Dunbar K Atallah H, Haight T, Vermetten E. Randomized Controlled Trial of Motion-Assisted Exposure Therapy for Posttraumatic Stress Disorder after Mild Traumatic Brain Injury, with and without an Eye Movement Task. Frontiers in Virtual Reality, 22 November 2022 https://doi.org/10.3389/frvir.2022.1005774.

DOCUMENTS (1):
  • Informed Consent Form (2019-10-10): https://cdn.clinicaltrials.gov/large-docs/36/NCT03796936/ICF_000.pdf